CLINICAL TRIAL: NCT01094951
Title: Engaging Depressed Low-Income Seniors in Mental Health Services
Acronym: ENGAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P30MH085943-03 (NIH); P30MH085943-03 (NIH); P30MH085943 (NIH)
Record Dates: First submitted 2010-03-26; First posted 2010-03-29 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Depression
Keywords: Depression
MeSH Terms: conditions — Depression | interventions — engage 8200

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ENGAGE (Other): In stage 1, study investigators will train Neighborhood House caseworkers to screen their clients for depressive symptoms.
  In stage 2, study investigators will train Neighborhood House caseworkers to use the ENGAGE intervention in referring their clients to mental health services
  Interventions: Behavioral: ENGAGE

INTERVENTIONS:
Behavioral: ENGAGE — During Stage 2, investigators will train Neighborhood House caseworkers to 1. provide psychoeducation that addresses client-specific barriers to evaluation and care; 2. use shared decision-making strategies to engage seniors and arrive at a decision about where and from whom to receive an evaluation and possible care; and 3. provide connections to preferred community-based mental health services.

SUMMARY:
This two-stage research study will

1. train caseworkers in three participating New York City Neighborhood Houses to screen their clients for depression, and
2. examine the usefulness of training these caseworkers in an intervention that targets barriers seniors face in receiving mental health services. In this intervention, called ENGAGE, Case Workers will: 1. identify and address seniors' barriers to receiving mental health services; 2. include the seniors' preferences in deciding which treatment options to choose; and 3. help seniors connect with affordable mental health services of their choice.

DETAILED DESCRIPTION:
In this research study, study investigators are partnering with United Neighborhood Houses of New York, the umbrella membership organization of the 34 New York City Neighborhood Houses. Due to the limited scope of this feasibility study, we have selected three Houses to serve as recruitment sites. These three house approximate the gender and racial characteristics of the larger group.

During Stage 1, investigators will work with the three Houses in implementing systematic research assessments to identify level of psychopathology, referral patterns, and connections to mental health evaluation among their depressed senior clients. Investigators will train caseworkers to screen their clients for depression and will also instruct caseworkers to refer any senior scoring endorsing depressive symptoms to their partnering community-based mental health or medical clinic. Data on successful connections to mental health evaluation will serve as the comparison to that achieved by Stage 2, the ENGAGE intervention.

During Stage 2 study investigators will train all caseworkers from each Neighborhood House to use the ENGAGE intervention. For eligible depressed seniors, the caseworker will:

1. provide psychoeducation that addresses client-specific barriers to evaluation and care (e.g., stigma, transportation);
2. use shared decision-making strategies to engage seniors and arrive at a decision about where and from whom to receive an evaluation and possible care; and
3. provide connections to preferred mental health services. Mental health service options will include referral to the senior's primary care physician or local community mental health clinic for further evaluation.

In two subsequent sessions 2 and 4 weeks later, the caseworker will assess success in receiving a mental health evaluation, and in initiating treatment:

* If the senior has not yet pursued an evaluation, the caseworker will continue to address his/her individual barriers and will re-engage in shared decision-making if necessary.
* If the senior did receive an evaluation that confirms a depressive diagnosis, but remains undecided about treatment, the case worker will empower and help the senior to select an appropriate treatment of his/her choice and will encourage ongoing engagement in this treatment.
* If an evaluation revealed the absence of a depressive disorder and no treatment recommendations, the caseworker will re-assess to ensure that depression did not emerge.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and older.
* Positive screen for major depression (PHQ-9 greater than 10): We chose standard PHQ-9 screening to correspond to routine procedures within each House that identify seniors in need of evaluation for treatment.
* Capacity to provide written consent for both research assessment and treatment. This criterion is necessary because subjects must be able to participate meaningfully in the interventions offered by the study and the assessment procedures.
* Working knowledge of English. Fluency in English sufficient for comprehending questionnaires of the study and/or for understanding the case worker. English does not have to be the subject's first language.

Exclusion Criteria:

* MMSE score < 24 or clinical diagnosis of dementia. Dementia, or cognitive impairment at this level may limit the senior's ability to participate in the intervention.
* Psychotic or manic symptoms or alcohol or substance dependence. These symptoms and disorders will be determined by the SCID assessment and require alternative interventions than those offered by the study. We focus in this project on seniors with depressive symptoms given existing Neighborhood House procedures for standard depression screening, and given difficulties in training case worker staff on screening for other psychiatric disorders. If this project is successful, we may then expand our efforts to target other disorders such as psychotic, manic, and alcohol and substance abuse and dependence disorders.
* Antidepressant medication or psychotherapy in the 4 weeks prior to baseline evaluation. The intervention is focused on linking depressed seniors who are in need of mental health services rather than those currently receiving treatment.
* Acute or severe medical illness: i.e., delirium, metastatic cancer, decompensated cardiac, liver or kidney failure, major surgery, stroke or myocardial infarction during the three months prior to entry; or drugs often causing depression, e.g., steroids, reserpine, alpha-methyl-dopa, tamoxifen, vincristine.
* Antisocial personality by DSM-IV: This disorder will possibly interfere with adherence to research procedures and treatment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of ENGAGE intervention | Measured at Baseline, 4, 8, and 12 weeks
  Examine the feasibility of training case workers in 3 Neighborhood Houses in ENGAGE - an intervention that identifies and addresses attitudinal and concrete barriers to pursuing evaluation and care; incorporates shared decision making in service and treatment options; and facilitates connection to affordable mental health services.

SECONDARY OUTCOMES:
Increase in referrals for mental health evaluation | Measured at Baseline, 4, 8, and 12 weeks
  Conduct a preliminary study to evaluate whether ENGAGE can increase the number of seniors (with symptoms of depression on a screen) who follow through with a referral for mental health evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Raue, Ph.D., Principal Investigator — Weill Medical College of Cornell University; George S. Alexopoulos, M.D., Study Director — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: No